CLINICAL TRIAL: NCT06607874
Title: Eligibility and Participation Characteristics of a Pilot Study of Self-Collection for Cervical Cancer Screening and HPV Vaccination for Cancer Prevention
Brief Title: Self-Collection for Cervical Cancer Screening and HPV Vaccination for Cancer Prevention Among Women in Emergency Care in Northeast Florida
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-009193; NCI-2024-07532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009193 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Human Papillomavirus-Related Cervical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observational aim 1 & aim 3: Patients may choose to undergo HPV vaginal swab self-collection on study in the research clinic or at home. Patients may choose to complete an interview on study. In addition, patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Observational aim 2: Patients are contacted by the study Clinical Research Coordinator (CRC) by phone on study and informed of HPV vaccination eligibility, asked interest in being vaccinated, and informed of sites for HPV vaccination. Patients are then contacted again by the CRC to determine if HPV vaccination occurred.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional study

SUMMARY:
Human Papilloma Virus (HPV) is a cause of cervical cancer in women. This study is being done to identify sites for cervical cancer screening and education regarding HPV vaccination outside of the traditional settings of primary care and gynecologic clinics. Identifying non-traditional cancer screening settings may increase cancer screening completion and HPV vaccination among women with limited health care knowledge and access who are vulnerable to health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Adults assigned as female at birth age 18-65 with a Mayo Clinic medical record number

Exclusion Criteria:

* Adults assigned as female at birth age 0-17
* Adults assigned as female at birth age > 65
* Adults assigned as male at birth
* Adults assigned as female at birth without a Mayo Clinic medical record number

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients recruited after previous ED visits
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Human Papilloma Virus (HPV) sample self-collection following Emergency Department (ED) presentation | Baseline
  Will be assessed by the percentage of women between 25-65 eligible for cervical cancer screening who participate or who opt not to participate in self-collection.
HPV vaccination following ED presentation | One month
  Will be assessed by the percentage of women between 18-26 eligible for HPV vaccination for cervical cancer prevention who participate in HPV vaccination. Participants will be contacted one month after initial contact to determine if the HPV vaccination was administered.
Interviews of women who decline self-collection | Baseline
  Phone or video-based interviews will be conducted with eligible participants who decline self-collection to determine reasons for non-participation.
Interviews of women who consent to self-collection but do not complete the self-collection | Up to 6 weeks
  Phone or video-based interviews will be conducted with participants who agree to participate but do not complete self-collection after 4 weeks to determine reasons for non-participation.
Interviews of women who complete the self-collection | Up to 6 weeks
  Phone or video-based interviews will be conducted with participants who completed self-collection for feedback on the process.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. DeStephano, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials